CLINICAL TRIAL: NCT06000904
Title: Evaluation and Improving Strategy of Turning Performance in Individuals With Stroke
Brief Title: Strategy of Turning Performance in Individuals With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU112118AF
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Turning performance; Balance performance; Exergame; Balance training; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame-based balance training group (Experimental)
  Interventions: Other: Exergame-based balance training
- Upper limb and trunk training group (Active Comparator)
  Interventions: Other: Upper limb and trunk training

INTERVENTIONS:
Other: Exergame-based balance training — For a four-week intervention consisting of three weekly sessions, each lasting 60 minutes. Each training session will include a 5-minute warm-up activity, 40-minute balance exercise, and 15-minute ground walking as a cool-down.
  Arms: Exergame-based balance training group
Other: Upper limb and trunk training — For a four-week intervention consisting of three weekly sessions, each lasting 60 minutes. Each training session will include a 5-minute warm-up activity, 40-minute upper-limb and trunk exercise, and 15-minute ground walking as a cool-down.
  Arms: Upper limb and trunk training group

SUMMARY:
This is a single-blind randomized controlled trial study. Thirty individuals with chronic stroke will be recruited and randomly assigned to the experimental and control groups. Subjects in the experimental group will receive exergame-based balance training, while subjects in the control group will receive upper limb and trunk training. Both groups will undergo a four-week intervention consisting of three sessions per week, each lasting 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* single incident of stroke
* stroke duration of at least 6 months
* lower limb Brunnstrom motor recovery stage between level three and five
* Functional Ambulation Categories scale ≥3

Exclusion Criteria:

* Individuals with cognitive impairmen (the Mini-Mental State Examination with a score below 24)
* visual or auditory impairments
* communication disorders
* other neurological diseases affecting motor performance, or any orthopedic conditions that could influence walking ability
* contraindications to physical activity, such as angina or uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Turning velocity (degrees/second) | Change from baseline at 4 weeks
Number of steps taken during turning | Change from baseline at 4 weeks
Turning step length (cm) | Change from baseline at 4 weeks
Stance phase duration (%) during turning | Change from baseline at 4 weeks
Swing phase duration (%) during turning | Change from baseline at 4 weeks

SECONDARY OUTCOMES:
Berg Balance Scale | Change from baseline at 4 weeks
  The Berg Balance Scale is employed to evaluate the functional balance ability of the subjects. This tool comprises 14 individual tests, each scored on a scale from 0 to 4, resulting in a total score of 56. A higher score indicates better balance ability.
Limits of stability test | Change from baseline at 4 weeks
  The limits of stability test is used to evaluate the dynamic balance ability of participants. Overall percentage is defined as the amount of direction control accuracy the individual has when performing the test. A higher percentage reflects better performance.
Modified clinical test of sensory interaction in balance | Change from baseline at 4 weeks
  This test is designed to assess sensory integration ability basing on the conditions of eyes open or closed and stable or unstable ground. The test is conducted in four contexts: context 1 involves standing with eyes open on a firm surface; context 2 involves standing with eyes open on a foam cushion; context 3 involves standing with eyes closed on a firm surface; and context 4 involves standing with eyes closed on a foam cushion. The overall sway index will be recorded for each condition of each trial, which will be summed the average of each condition.
Walking velocity (cm/sec) in straight walk | Change from baseline at 4 weeks
Step length (cm) in straight walk | Change from baseline at 4 weeks
Cadence (steps/minute) in straight walk | Change from baseline at 4 weeks
Stance phase duration (%) in straight walk | Change from baseline at 4 weeks
Swing phase duration (%) in straight walk | Change from baseline at 4 weeks
Time Up and Go test | Change from baseline at 4 weeks
  The Timed Up & Go (TUG) test is employed to evaluate the activity functionality of participants. The average time taken for completion will be recorded for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided